CLINICAL TRIAL: NCT07349303
Title: Neoadjuvant Pembrolizumab in Patients With Stage IIb/c Melanoma, a Phase II Double-blind Placebo-controlled Randomized Trial
Brief Title: Neoadjuvant Pembrolizumab in Patients With Stage IIb/c Melanoma
Acronym: NEOPRIME
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-519594-19-00; 2024-519594-19-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Melanoma (Skin Cancer)
Keywords: IMMUNOTHERAPY; PRIMARY CUTANOUS MELANOMA; NEOPRIME trial; NEOADJUVANT TREATMENT
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab (Experimental): Patients will receive one dose of intravenous pembrolizumab and then 4 weeks later undergo WLE and SLNB.
  Interventions: Drug: Pembrolizumab
- Placebo (Placebo Comparator): Patients will receive one dose of intravenous placebo and then 4 weeks later undergo WLE and SLNB.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pembrolizumab — Immunotherapy
  Arms: Pembrolizumab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A phase II double-blind placebo-controlled randomized trial. Patients with a clinical suspicion of a thick primary melanoma without clinical suspicion or evidence of lymph-node engagement will undergo a 3 mm punch biopsy to verify the diagnosis and ascertain eligibility. Patients will receive 1 cycle of pembrolizumab 400 mg or placebo and 4 weeks later undergo a wide local excision and sentinel lymph node biopsy according to the national guideline recommendations .

The primary objective is to evaluate the pathological response of one cycle of neoadjuvant pembrolizumab in patients with biopsy-proven stage IIb/c melanoma. Secondary objectives include efficacy and safety analysis, as well as biomarker discovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years.
2. Signed informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
4. Histopathologically confirmed primary cutaneous melanoma stage IIb/c (Breslow >2.0 mm with ulceration OR Breslow >4.0mm without ulceration) with a minimum diameter of 5 mm not completely removed by the diagnostic biopsy
5. Patient planned for wide local excision and sentinel lymph node biopsy
6. Adequate organ function on blood test
7. Female patient of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female patients of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 150 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
9. Male patients of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 150 days after the last dose of study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Life expectancy of less than 3 years.
2. Patients who are unable to undergo general anesthesia for any reason.
3. Clinical or radiographic evidence of nodal, satellite, in-transit or distant metastases
4. Risk for developing in-operable disease due to study procedures as judged by study investigator
5. Prior immunotherapy for any malignancy
6. Use of live vaccines four weeks before or after the last study treatment.
7. History of severe reactions to monoclonal antibodies.
8. Active autoimmune disease or a documented history of autoimmune disease requiring systemic immunomodulatory treatment. Diabetes, rheumatoid arthritis, psoriasis, atopic dermatitis and hypothyroidism are excepted.
9. A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
10. Concomitant therapy with any other anti-cancer therapy, concurrent medical conditions requiring use of immunosuppressive medications or use of other investigational drugs.
11. Has a known additional malignancy that is progressing or requires active treatment.
12. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 150 days after the last dose of study drug.
13. A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-05-15 (Estimated); Study Completion 2031-05-15 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | 48 month
  Pathological response rate in the primary tumor according to adapted guidelines of the International Neoadjuvant Consortium (14)
  The pathological response will be described:
  * Complete pathological response (pCR) - 0% viable tumor cells in the surgical specimen
  * Near complete pathological response (near pCR) - ≤10% viable tumor
  * Partial pathological response (pPR) - >10%-≤50% viable tumor
  * No pathological response (pNR) - >50% viable tumor The proportion of patients with a pCR, near pCR or pPR will determine the pathological response rate.

SECONDARY OUTCOMES:
Frequency and severity of adverse events (AEs) and serious adverse events (SAEs) | 48 month
  The proportion of patients with adverse events (AE) as described in CTCAE version 5.0, from the initiation of study treatment until 100 days after the end of treatment:
  1. Proportion of patients with an AE by CTCAE term and grade.
  2. Proportion of patients with grade 3/4 AEs by AE term.
  3. The duration of events reported in (a)
  4. Proportion of patients with requirement to delay surgery due to an AE.
  5. Proportion of patients with a requirement to permanently discontinue study treatment due to an AE.
  6. The proportion of patients with a requirement for oral or parenteral steroid treatment for immunology-related adverse events.
  7. The proportion of patients with post-operative complications (e.g. seroma formation, wound infection or lymphoedema) and duration of events.
Feasibility of neoadjuvant therapy in stage II melanoma | 48 month
  1. Proportion of eligible patients who consent to the study.
  2. Proportion of included patients who complete all treatment according to protocol.
Sentinel lymph node positivity rate | 48 month
  1. The proportion of patients undergoing a sentinel node biopsy who have a positive result in the lymph node.
  2. The number of sentinel nodes identified and the number harvested.
  3. The proportion of patients with a positive sentinel node biopsy who undergo completion lymph node dissection.
Local recurrence rate | 48 month
  The proportion of patients after surgery with histologically confirmed diagnosis of local disease recurrence, as detected by the patient, on physical examination or during imaging surveillance.
Regional recurrence rate | 48 month
  The proportion of patients after surgery with histologically confirmed diagnosis of regional disease recurrence, as detected by the patient, on physical examination or during imaging surveillance
Event free survival (EFS) | 48 month
  The proportion of patients that did not undergo surgery or histologically confirmed diagnosis of disease recurrence (local, regional, and distant), as detected by the patient, on physical examination or during imaging surveillance, or death from any cause.
To assess recurrence free survival (RFS). | 48 month
  The proportion of patients after surgery with histologically confirmed diagnosis of disease recurrence (local, regional, and distant), as detected by the patient, on physical examination or during imaging surveillance, or death from any cause.
Distant metastasis-free survival (DMFS) | 48 month
  The proportion of patients after surgery with histologically confirmed diagnosis of disease distant recurrence, as detected by the patient, on physical examination or during imaging surveillance, or death from any cause.
Melanoma specific survival (MSS) | 48 month
  The proportion of patients who die, from the initiation of study treatment to the date of death from melanoma.
Overall survival (OS) | 48 month
  The proportion of patients who die, from the initiation of study treatment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No